CLINICAL TRIAL: NCT01190007
Title: A Multi-Center, Open Label Study To Evaluate Long Term Safety Of Caduet In Patient With Both Of Hypertension And Hypercholesterolemia, Or With Both Of Angina Pectoris And Hypercholesterolemia
Brief Title: Open Label Study To Evaluate The Long-Term Safety Profiles Of Caduet In Japanese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3841064
Record Dates: First submitted 2010-08-05; First posted 2010-08-27 (Estimated); Results first posted 2012-12-03 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Hypertension; Hypercholesterolemia; Angina Pectoris
MeSH Terms: conditions — Hypertension; Hypercholesterolemia; Angina Pectoris | interventions — amlodipine, atorvastatin drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caduet (Experimental)
  Interventions: Drug: Caduet

INTERVENTIONS:
Drug: Caduet — One Caduet tablet will be administered once daily after breakfast, in principle, for 52 weeks

SUMMARY:
The primary objective is to investigate the safety of Caduet (2.5 mg/5 mg, 2.5 mg/10 mg, 5 mg/5 mg or 5 mg/10 mg as dose of Amlodipine/Atorvastatin) during 52 weeks treatment period in Japanese patients with both of hypertension and hypercholesterolemia, or with both angina pectoris and hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Subject with both hypertension and hypercholesterolemia must meet the following (1), and the following (2) or (3):
* (1) Subjects who take Amlodipine 2.5mg/day or 5mg/day at least 28 days before Week -2, and Subjects with well controlled BP value (BP value < 140/90mmHg at Week 0)
* (2) Subjects who take Atorvastatine 5mg/day or 10mg/day at least 28days before Week -2
* (3) Statin-naïve patient, defined as receiving no statin therapy for more than 3 months during the previous 12 months, with LDL-C ≥ 160 mg/dL, LDL-C < 250 mg/dL, and TG < 400 mg/dL at Week -2
* Subject with both angina pectoris and hypercholesterolemia must meet the following (1), and the following (2) or (3):
* (1) Subjects who take Amlodipine 2.5mg/day or 5mg/day at least 28 days before Week -2, and who meet the following criteria; Subjects with well controlled BP value (BP value < 140/90mmHg at Week 0), and subjects with clinically stable of angina pectoris
* (2) Subjects who take Atorvastatine 5mg/day or 10mg/day at least 28days before Week -2
* (3) Statin-naïve patient, defined as receiving no statin therapy for more than 3 months during the previous 12 months, with LDL-C ≥ 160 mg/dL, LDL-C < 250 mg/dL, and TG < 400 mg/dL at Week -2

Exclusion Criteria:

* Subjects who need three or more multi-antihypertensive therapies to achieve the target BP level or uncontrolled status of hypertension at Week 0 (V1); the target BP level is defined as systolic blood pressure < 140mmHg and diastolic blood pressure < 90 mmHg.
* Uncontrolled or uncontrollable status of hypercholesterolemia at Week -2; A LDL-C ≥ 160 mg/dL even though Atorvastatine 10 mg has administrated

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2010-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- Japan (20):
  - Healthcare Corporation MEDOC Medical Dock&Clinic, Nagoya, Aichi-ken
  - Beppu Medical Clinic, Dazaifu, Fukuoka
  - Morizono medical clinic, Kitakyushu, Fukuoka
  - Gakkentoshi Clinic, Nishiku, Fukuoka
  - Department of internal gastro-intestinal medicine Ohshima clinic, Sapporo, Hokkaido
  - Oofuji Clinic, Amagasaki, Hyōgo
  - Mizutani Clinic, Kobe, Hyōgo
  - Nada Clinic, Kobe, Hyōgo
  - Idaimae-naika Clinic, Kawasaki, Kanagawa
  - Sakakibara Clinic, Wakaumekai Medical Corporation, Yokohama, Kanagawa
  - Masunaga Clinic, Fujimi, Saitama
  - Sugiura Clinic, Kawaguchi, Saitama
  - Masuda Clinic, Adachi-ku, Tokyo
  - Wakasugi Family Clinic, Arakawa-ku, Tokyo
  - Medical Care Law Person Corporation Kenseikai, Kobayashi Internal Medicine Clinic, Koto-ku, Tokyo
  - Banno Clinic, Ohta-ku, Tokyo
  - Hatano Medical Clinic, Setagaya-ku, Tokyo
  - Suzuki Circulatory Medical Clinic, Setagaya-ku, Tokyo
  - Yano Cardiovascular Clinic, Fukuoka
  - Nakaoka Clinic, Osaka

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3841064&StudyName=Open%20Label%20Study%20To%20Evaluate%20The%20Long-Term%20Safety%20Profiles%20Of%20Caduet%20In%20Japanese%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Caduet: Single pill combination of amlodipine and atorvastatin (Caduet) of the specified strength (2.5 mg/5 mg, 2.5 mg/10 mg, 5 mg/5 mg, or 5 mg/10 mg, as Amlodipine/Atorvastatin) was administered once daily for 52 weeks. Caduet doses were determined according to the doses of amlodipine and atorvastatin which were administered prior to the study assignment in line with the levels of blood pressure and low-density lipoprotein cholesterol (LDL-C) at Week 0. The fixed dose was administered up to Week 12, then, the dose was adjusted based on the blood pressure and LDL-C observed after.
Period: Overall Study
Arm/Group | Caduet
Started | 159 (Treated)
Completed | 145
Not Completed | 14
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 8
Not completed — Difficulty of visit for complications | 1
Not completed — Participant was arrested | 1

BASELINE CHARACTERISTICS:
Arm/Group | Caduet
Number analyzed (Participants) | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Relatedness to [study drug] was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Time Frame: 52 weeks
Population: The safety analysis set included all participants who took at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Caduet
Number analyzed (Participants) | 159
Participants
  AE | 120
  SAE | 11

2. Secondary Outcome: Change From Baseline in Trough Systolic Blood Pressure (SBP) at Each Visit in Participant Population With Both Hypertension and Hypercholesterolemia
Description: Value at each visits minus value at baseline
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: The efficacy analysis set included all participants who took at least one dose of study drug and contributed data to baseline and at least one post-baseline efficacy assessment. LOCF means Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Caduet
Number analyzed (Participants) | 142
mmHg
  Week 2 (n=140) | -0.2 (8.57)
  Week 4 (n=139) | -0.6 (9.19)
  Week 8 (n=140) | 0.0 (10.38)
  Week 12 (n=140) | -0.4 (10.46)
  Week 16 (n=138) | -1.5 (11.10)
  Week 20 (n=136) | -2.8 (10.07)
  Week 24 (n=134) | -1.8 (9.74)
  Week 28 (n=132) | -3.1 (10.39)
  Week 32 (n=132) | -4.8 (10.76)
  Week 36 (n=132) | -4.8 (8.85)
  Week 40 (n=132) | -4.4 (8.84)
  Week 44 (n=130) | -4.0 (10.58)
  Week 48 (n=130) | -2.3 (10.20)
  Week 52 (n=129) | -1.5 (10.92)
  Week 52 (LOCF) (n=142) | -1.5 (10.81)

3. Secondary Outcome: Change From Baseline in Trough Systolic Blood Pressure (SBP) at Each Visit in Population With Both Angina Pectoris and Hypercholesterolemia
Description: Value at each visits minus value at baseline
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: The efficacy analysis set included all participants who took at least one dose of study drug and contributed data to baseline and at least one post-baseline efficacy assessment. Participants both angina pectoris and hypercholesterolemia were included the participants with all of angina pectoris, hypertension and hypercholesterolemia.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Caduet
Number analyzed (Participants) | 16
mmHg
  Week 2 (n=15) | -1.1 (11.57)
  Week 4 (n=16) | -2.3 (8.68)
  Week 8 (n=16) | -1.1 (7.76)
  Week 12 (n=16) | -2.2 (9.11)
  Week 16 (n=16) | -2.3 (13.49)
  Week 20 (n=16) | -2.3 (8.47)
  Week 24 (n=16) | -6.7 (9.07)
  Week 28 (n=16) | -6.8 (10.23)
  Week 32 (n=16) | -7.8 (10.79)
  Week 36 (n=15) | -5.7 (9.72)
  Week 40 (n=15) | -2.7 (10.00)
  Week 44 (n=15) | -3.7 (11.38)
  Week 48 (n=15) | -0.4 (9.44)
  Week 52 (n=15) | -4.4 (13.08)
  Week 52 (LOCF) (n=16) | -3.1 (13.77)

4. Secondary Outcome: Change From Baseline in Trough Diastolic Blood Pressure (DBP) at Each Visit in Participant Population With Both Hypertension and Hypercholesterolemia
Description: Value at each visits minus value at baseline
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Caduet
Number analyzed (Participants) | 142
mmHg
  Week 2 (n=140) | 0.3 (7.03)
  Week 4 (n=139) | -0.4 (6.75)
  Week 8 (n=140) | 0.2 (6.90)
  Week 12 (n=140) | -0.2 (7.13)
  Week 16 (n=138) | -0.7 (7.50)
  Week 20 (n=136) | -1.8 (7.38)
  Week 24 (n=134) | -1.6 (7.03)
  Week 28 (n=132) | -2.6 (7.27)
  Week 32 (n=132) | -3.5 (7.84)
  Week 36 (n=132) | -4.3 (6.50)
  Week 40 (n=132) | -3.2 (6.90)
  Week 44 (n=130) | -2.5 (7.40)
  Week 48 (n=130) | -2.0 (7.52)
  Week 52 (n=129) | -0.6 (7.72)
  Week 52 (LOCF) (n=142) | -0.6 (7.68)

5. Secondary Outcome: Change From Baseline in Trough Diastolic Blood Pressure (DBP) at Each Visit in Participant Population With Angina Pectoris and Hypercholesterolemia
Description: Value at each visits minus value at baseline
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: The efficacy analysis set included all participants who took at least one dose of study drug and contributed data to baseline and at least one post-baseline efficacy assessment.
  Participants with both angina pectoris and hypercholesterolemia were included the participants with all of angina pectoris, hypertension and hypercholesterolemia.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Caduet
Number analyzed (Participants) | 16
mmHg
  Week 2 (n=15) | 0.8 (8.21)
  Week 4 (n=16) | -1.1 (4.96)
  Week 8 (n=16) | -1.0 (6.19)
  Week 12 (n=16) | -1.1 (6.86)
  Week 16 (n=16) | -2.2 (7.12)
  Week 20 (n=16) | -0.9 (6.71)
  Week 24 (n=16) | -3.5 (6.69)
  Week 28 (n=16) | -3.0 (6.55)
  Week 32 (n=16) | -4.8 (9.56)
  Week 36 (n=15) | -2.5 (6.20)
  Week 40 (n=15) | -1.2 (8.53)
  Week 44 (n=15) | -2.6 (9.06)
  Week 48 (n=15) | -0.7 (5.18)
  Week 52 (n=15) | -4.4 (6.75)
  Week 52 (LOCF) (n=16) | -3.2 (8.29)

6. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) at Each Visit
Description: "Value at each visits minus value at baseline" divided by value at baseline multiplied by 100
Time Frame: Weeks 4, 12, 24, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of LDL-C
Arm/Group | Caduet
Number analyzed (Participants) | 157
Percentage of LDL-C
  Week 4 (n=157) | -10.9 (23.87)
  Week 12 (n=155) | -7.4 (25.66)
  Week 24 (n=151) | -10.5 (24.04)
  Week 52 (n=144) | -12.3 (23.62)
  Week 52 (LOCF) (n=156) | -12.2 (23.55)

7. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC) at Each Visit
Description: "Value at each visits minus value at baseline" divided by value at baseline multiplied by 100
Time Frame: Weeks 4, 12, 24, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of TC
Arm/Group | Caduet
Number analyzed (Participants) | 157
Percentage of TC
  Week 4 (n=157) | -7.3 (15.90)
  Week 12 (n=156) | -5.0 (17.03)
  Week 24 (n=151) | -7.9 (16.78)
  Week 52 (n=145) | -8.0 (16.37)
  Week 52 (LOCF) (n=157) | -8.1 (16.04)

8. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) at Each Visit
Description: "Value at each visits minus value at baseline" divided by value at baseline multiplied by 100
Time Frame: Weeks 4, 12, 24, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of HDL-C
Arm/Group | Caduet
Number analyzed (Participants) | 157
Percentage of HDL-C
  Week 4 (n=157) | 1.5 (10.63)
  Week 12 (n=156) | 4.0 (13.91)
  Week 24 (n=151) | -0.5 (13.26)
  Week 52 (n=145) | 2.2 (11.47)
  Week 52 (LOCF) (n=157) | 2.5 (11.69)

9. Secondary Outcome: Percent Change From Baseline in Triglyceride (TG) at Each Visit
Description: "Value at each visits minus value at baseline" divided by value at baseline multiplied by 100
Time Frame: Week 4, 12, 24, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of TG
Arm/Group | Caduet
Number analyzed (Participants) | 157
Percentage of TG
  Week 4 (n=157) | 8.2 (52.47)
  Week 12 (n=156) | 3.6 (49.94)
  Week 24 (n=151) | 6.4 (45.75)
  Week 52 (n=145) | 8.5 (62.03)
  Week 52 (LOCF) (n=157) | 7.2 (60.92)

10. Secondary Outcome: Change From Baseline in Ratio of Low Density Lipoprotein Cholesterol (LDL-C) to High Density Lipoprotein Cholesterol (HDL-C) at Each Visit
Description: Value at each visits minus value at baseline
Time Frame: Weeks 4, 12, 24, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Caduet
Number analyzed (Participants) | 157
Ratio
  Week 4 (n=157) | -0.4 (0.70)
  Week 12 (n=155) | -0.3 (0.70)
  Week 24 (n=151) | -0.3 (0.66)
  Week 52 (n=144) | -0.4 (0.68)
  Week 52 (LOCF) (n=156) | -0.4 (0.68)

11. Secondary Outcome: Change From Baseline in Ratio of Total Cholesterol (TC) to High Density Lipoprotein Cholesterol (HDL-C) at Each Visit
Description: Value at each visits minus value at baseline
Time Frame: Weeks 4, 12, 24, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Caduet
Number analyzed (Participants) | 157
Ratio
  Week 4 (n=157) | -0.4 (0.77)
  Week 12 (n=156) | -0.4 (0.79)
  Week 24 (n=151) | -0.3 (0.76)
  Week 52 (n=145) | -0.4 (0.77)
  Week 52 (LOCF) (n=157) | -0.4 (0.77)

12. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Each Visit
Description: "Value at each visits minus value at baseline" divided by value at baseline multiplied by 100
Time Frame: Week 4, 12, 24, and 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of Apolipoprotein B
Arm/Group | Caduet
Number analyzed (Participants) | 157
Percentage of Apolipoprotein B
  Week 4 (n=157) | -9.2 (18.59)
  Week 12 (n=156) | -5.8 (21.13)
  Week 24 (n=151) | -7.4 (20.99)
  Week 52 (n=145) | -9.1 (20.10)
  Week 52 (LOCF) (n=157) | -9.3 (19.84)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Caduet
Serious Adverse Events (participants affected / at risk) | 11/159
Other Adverse Events (participants affected / at risk) | 101/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caduet (N=159)
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aortic aneurysm (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Caduet (N=159)
Abdominal discomfort (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 5
Gastritis (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5
Bronchitis (Infections and infestations) | 11
Cystitis (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 53
Pharyngitis (Infections and infestations) | 17
Fall (Injury, poisoning and procedural complications) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4
Periarthritis (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 6
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 8
Eczema (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.